CLINICAL TRIAL: NCT04007861
Title: Exploring the Link Between Cancer Genetics and Persistent Post-surgical Pain (PPSP) Following Breast Cancer Treatment
Brief Title: Exploring the Link Between Cancer Genetics and PPSP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5006
Record Dates: First submitted 2019-06-21; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Cancer-related Pain; Chronic Post Cancer Surgery Pain; Breast Cancer
MeSH Terms: conditions — Cancer Pain; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pain: This will be the group of patients in whom pain is a significant enough problem, that they have been referred to the specialist Pain Management Team. These patients will be identified retrospectively.
  Patients seen in Pain Management Clinics between 1st of January 2016 and 31st of December 2018, who have consented to be included in the Pain Management database and have a clinician specified pain diagnosis of pain persistent post-surgical pain following breast cancer treatment will be identified. If these patients have an unclear pain diagnosis, they will not be included.
- Patients without pain: This will be the group of patients in whom pain is deemed not to be a significant problem.
  Once again, these patients will be identified retrospectively. Appropriately matched patients to the 52 patients in the "patients with pain" will be identified using records of hospital operating lists by the peri-operative medicine team.
  Patients will be matched based upon the following details:
  * Age (within 5 years of matched case)
  * Surgical procedure (matched for the following elements:
    * Surgery to breast tissue (biopsy, lumpectomy, wide-local excision or mastectomy)
    * +/- Sentinal lymph node biopsy or axillary dissection
    * +/- Reconstruction
  * Surgical procedure within 3-months of matched case.
  Provided these individuals have not had an appointment with or referral to the Pain Management Team, they will be included in the matched controls.

SUMMARY:
Pain is common in cancer, affecting between 40 and 60% of patients depending on tumour type and stage of disease, and represents a major area of unmet need in cancer survivors. Despite advances in treatment, there has been no significant reduction in those who experience pain. Breast cancer is common. It represents 10% of newly diagnosed cancers globally and is often associated with pain.

Exact physiological mechanisms for cancer pain are not yet fully established. There is a complex relationship between a malignant lesion and its micro-environment; a tumour does not exist in isolation but has a dynamic relationship with host cells. There is a growing interest in delineating the relationship between tumour manifestations and pain.

By retrospectively identifying individuals who have been referred to specialist pain clinics at a cancer centre and matching them to controls, the investigators can identify two groups of patients (those who experienced significant problems with pain and those who did not). Accessing paraffin-embedded tissue samples from those that have had surgical resections, will allow the investigators to compare tissue samples, in particular the metabolic and genetic differences, between the two groups.

No new tissue samples will be required for this study.

Pain is a major area of unmet need in cancer survivors. The investigators propose that this project would provide valuable knowledge and pilot data regarding the link between pain and tumour genetics. It has the potential to identify tumour genes or mutations that are associated with greater incidences of pain and ultimately potentially guide targeted interventions to help reduce the frequency and impact of pain on patients living with and beyond cancer.

DETAILED DESCRIPTION:
This study will be a retrospective, case-control study. There will be two groups of patients identified retrospectively:

The first group will be patients who have been referred to the pain management team for persistent-post surgical pain following breast cancer treatment.

The second group, will consist of patients who have been matched for age, procedure and time-lapsed since operation. These patients will not have persistent post-surgical pain.

Archived paraffin-embedded tissue samples, that have previously been taken from these patients, will be required. Samples accessed will be from patients who have previously provided consent for their samples to be used for research purposes. Once appropriate samples have been identified by the tissue banks, all data will be pseudonymised. This will include details that patients have consented to providing for research purposes via the Pain Management Database, which has Trust (CCR 442) and Research Ethics Committee (REC 16/LO/1989) approval.

Laboratory studies will then be conducted to A) investigate the underlying variations of the PIK3CA gene of tumours within the two cohorts of patients, B) investigate other genetic variations between these two groups and C) establish the key genetic and signalling pathway alterations between these two groups.

The methods by which these investigations will be conducted will be by performing PIK3CA genomics, genetic profiling, next generation sequencing and finally immunohistochemistry for activation of signalling pathways.

This study will analyse archived paraffin embedded tissue samples in a laboratory only.

The anticipated time-scale for this project would be approximately one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving treatment at the Royal Marsden Hospital.
* Patients with a diagnosis of primary breast cancer.
* Patients who have had surgical resection of their breast tumour.
* Paraffin-embedded tissue samples available from Royal Marsden Tissue Banks.

Exclusion Criteria:

* Under 18 years of age.
* Lack of adequate tissue sample available from the Tissue Bank.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Although two groups of patients will be identified retrospectively:
  1. The first group will be patients who have been referred to the pain management team for persistent-post surgical pain following breast cancer treatment.
  2. The second group, will consist of patients who have been matched for age, procedure and time-lapsed since operation. These patients will not have persistent post-surgical pain.
  Ultimately, archived paraffin-embedded tissue samples, that have previously been taken from these patients, will be requested. Samples accessed will be from patients who have previously provided consent for their samples to be used for research purposes.
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of mutations of the PIK3CA gene. | Within 6-8months
  PIK3CA genomics will result in a binary measure (either wild-type or mutant). The difference in proportion of the PIK3CA gene mutation in those with persistent post-surgical pain compared with those without persistent post-surgical pain will be the primary outcome measure.

SECONDARY OUTCOMES:
Proportion of individual gene mutations in pain group compared with the no pain group. | Within 6-8months
  DNA analysis will determine the presence or absence of other gene mutations (binary outcome).
Difference in mean gene expression in those with pain compared with those without pain. | Within 6-8months
  Exploring the difference in gene expression between the two groups.
Proportion of individual DNA copy number changes (either amplification/gain or loss) in those with pain compared with those without pain. | Within 6-8months
  DNA copy number can either be unchanged or changed. Changes are described as either 'amplification/gain' or 'loss'. Data will be analysed as binary data (either no change or change).
Frequency of changes to DNA copy number (either amplification/gain or loss) in those with pain compared with those without pain. | Within 6-8months
  DNA copy number can either be unchanged or changed. Changes are described as either 'amplification/gain' or 'loss'. Data will be analysed as binary data (either no change or change).
Difference in median of magnitude of activation status of signalling pathways between those with pain and those without pain. | Within 6-8months
  Comparison the activation status of signalling pathways between the two groups. The magnitude of activation status will be reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Brown, MBBS, Principal Investigator — Royal Marsden NHS Foundation Trust